CLINICAL TRIAL: NCT03931746
Title: Porcine Xenograft Versus Second Intention Healing: a Randomized, Evaluator-blinded Clinical Trial
Brief Title: Porcine Xenograft Versus Second Intention Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company discontinued production of the Porcine Xenograft
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Victoria Sharon, Director - Dermatologic Surgery & Dermato-Oncoly, Department of Dermatology, North Shore University Hospital, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0715
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Wound Healing and Scar Quality Following Mohs Surgery and Excisional Dermatologic Surgery

STUDY DESIGN:
Intervention Model Description: To compare wound healing and scar quality following the placement of a porcine xenograft compared to second intention healing of leg wounds following Mohs or excisional surgery.
Who Masked: Outcomes Assessor
Masking Description: The evaluator will not have knowledge of or access to the intervention that was performed and represents a provider not involved in the surgical care of the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Porcine Xenograft placement (Experimental): Porcine xenograft will be placed on the wound.
  Interventions: Device: Porcine xenograft
- No porcine xenograft (No Intervention): The wound will be allowed to heal via second intention.

INTERVENTIONS:
Device: Porcine xenograft — The EZ-DERM™ porcine xenograft is a biosynthetic dressing made from porcine collagen containing aldehyde crosslinking. It has been most commonly applied to the management of 2nd degree burns, both partial-thickness and full-thickness defects. This dressing can be used for two healing purposes, either for primary healing or as an intermediate in the preparation for a skin graft
  Arms: Porcine Xenograft placement

SUMMARY:
The purpose of this research study is to test whether it is better to allow patients with post- operative wounds on the legs to heal on their own without a covering or to use a porcine xenograft (skin graft that is made from pig cells) to cover the wound during healing. It is currently not known which option is better in terms of the appearance, complication rate or the impact on the patient's quality of life during the healing process. In this location, it is common receive either treatment.

DETAILED DESCRIPTION:
Porcine xenograft has been used as a barrier to the skin for over 30 years, and due to its wound healing promoting factors, we believe that its use may result in decreased healing time, smaller scar size, better cosmetic outcomes, lower pain levels, and decreased rates of infection and other post-surgical complications.

Upon completion of dermatologic surgery following standard procedures, patients will be randomized into one of two groups (porcine xenograft placement or second intention healing). Weekly follow-up via questionnaires will be conducted as well as a final office visit follow-up at 3 months.

The application of porcine xenograft dressings for wound healing was first studied in 1985, with evidence supporting several benefits when compared to traditional dressings [1]. Subsequent studies have substantiated the use of this dressing for a variety of clinical settings [2,3].

The EZ-DERM™ porcine xenograft is a biosynthetic dressing made from porcine collagen containing aldehyde crosslinking [1,3]. It has been most commonly applied to the management of 2nd degree burns, both partial-thickness and full-thickness defects [4]. This dressing can be used for two healing purposes, either for primary healing or as an intermediate in the preparation for a skin graft [2].

Compared to other biosynthetic dressings, porcine xenografts afford longer wound adherence and can be stored at room temperature [1]. The xenograft triggers rejection by the surgical defect, increasing local vascularization [5]. It also allows for rapid granulation, a reduced risk of infection, as well as reduced wound-related fluid and thermal losses [6-8]. There is also evidence that the quicker wound healing reduces the frequency of dressings, hospitalization time, pain, and analgesic [9,10].

Several clinical case series have extended the use of porcine xenografts to Mohs Micrographic Surgery (MMS) to facilitate post-operative wound care. Porcine xenograft dressings were determined to be safe, well-tolerated, and able to be applied to a wide anatomical range [3,12].

In addition to biosynthetic dressings, healing via second intention remains an alternative [13,14]. The extremities of elderly patients are a common location for wound granulation. Drawbacks to second intention healing on the extremities include prolonged healing time and extended wound care for the patient [15].

Chern et. al. completed a review of biological dressings in dermatologic surgery and concluded that there is a limited number of studies focusing on the conclusive benefits of dressings [16]. Although studies have established that EZ-DERM™ was helpful for wound healing following Mohs surgery, there have not been any definitive statistical measures reported in the literature. Additionally, there is a lack of studies assessing the direct comparison to second intention healing.

Our plan is to perform a direct comparison of porcine xenograft placement to second intent healing. Based on the previously studied benefits of the xenograft as a barrier to the skin and one which has wound healing promoting factors, we believe that its use may result in decreased healing time, smaller scar size, better cosmetic outcomes, lower pain levels, and decreased rates of infection and other post-surgical complications.

Our study will allow surgeons to make informed decisions on whether porcine xenograft dressing is superior to that of second intention healing and thus worth considering.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to give informed consent themselves
* Willing to return for follow-up visits
* Post-operative defects greater than 8 mm (in greatest diameter or length of circular or oval geometric shape) on the lower extremities (including the feet)
* Single defect

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Unwilling to return for follow-up
* Pregnant women
* Wounds less than 8 mm in length
* Wounds on the head, neck or digits
* Patients in which primary linear closure is recommended

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Sharon, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Northwell Health Physician Partners Division of Dermatology, Bay Shore, New York
  - Northwell Health Physician Partners Division of Dermatology, Lake Success, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanstraelen P. Comparison of calcium sodium alginate (KALTOSTAT) and porcine xenograft (E-Z DERM) in the healing of split-thickness skin graft donor sites. Burns. 1992 Apr;18(2):145-8. doi: 10.1016/0305-4179(92)90014-l. PMID 1590931
- [Background] Duteille F, Perrot P. Management of 2nd-degree facial burns using the Versajet((R)) hydrosurgery system and xenograft: a prospective evaluation of 20 cases. Burns. 2012 Aug;38(5):724-9. doi: 10.1016/j.burns.2011.12.008. Epub 2012 Feb 22. PMID 22360953
- [Background] Raimer DW, Group AR, Petitt MS, Nosrati N, Yamazaki ML, Davis NA, Kelly BC, Gibson BR, Montilla RD, Wagner RF Jr. Porcine xenograft biosynthetic wound dressings for the management of postoperative Mohs wounds. Dermatol Online J. 2011 Sep 15;17(9):1. PMID 21971266
- [Background] Chiu T, Burd A. "Xenograft" dressing in the treatment of burns. Clin Dermatol. 2005 Jul-Aug;23(4):419-23. doi: 10.1016/j.clindermatol.2004.07.027. PMID 16023938
- [Background] Demling RH, DeSanti L. Management of partial thickness facial burns (comparison of topical antibiotics and bio-engineered skin substitutes). Burns. 1999 May;25(3):256-61. doi: 10.1016/s0305-4179(98)00165-x. PMID 10323611
- [Background] Gerding RL, Imbembo AL, Fratianne RB. Biosynthetic skin substitute vs. 1% silver sulfadiazine for treatment of inpatient partial-thickness thermal burns. J Trauma. 1988 Aug;28(8):1265-9. doi: 10.1097/00005373-198808000-00022. PMID 3411648
- [Background] Hansbrough JF, Zapata-Sirvent R, Carroll WJ, Dominic WJ, Wang XW, Wakimoto A. Clinical experience with Biobrane biosynthetic dressing in the treatment of partial thickness burns. Burns Incl Therm Inj. 1984 Aug;10(6):415-9. doi: 10.1016/0305-4179(84)90081-0. PMID 6478287
- [Background] Horch RE, Jeschke MG, Spilker G, Herndon DN, Kopp J. Treatment of second degree facial burns with allografts--preliminary results. Burns. 2005 Aug;31(5):597-602. doi: 10.1016/j.burns.2005.01.011. Epub 2005 Mar 21. PMID 15993304
- [Background] Becker D. [Temporary dressing of burn wounds using sterile frozen porcine skin (author's transl)]. Unfallheilkunde. 1981 Apr;84(4):158-60. No abstract available. German. PMID 7233629
- [Background] Hosseini SN, Mousavinasab SN, Fallahnezhat M. Xenoderm dressing in the treatment of second degree burns. Burns. 2007 Sep;33(6):776-81. doi: 10.1016/j.burns.2006.10.396. Epub 2007 May 23. PMID 17524562
- [Background] Yang YW, Ochoa SA. Use of Porcine Xenografts in Dermatology Surgery: The Mayo Clinic Experience. Dermatol Surg. 2016 Aug;42(8):985-91. doi: 10.1097/DSS.0000000000000804. PMID 27340740
- [Background] Diwan R, Tromovitch TA, Glogau RG, Stegman SJ. Secondary intention healing. The primary approach for management of selected wounds. Arch Otolaryngol Head Neck Surg. 1989 Oct;115(10):1248-9. doi: 10.1001/archotol.1989.01860340102027. PMID 2789782
- [Background] Howe NR, Lang PG Jr. Daily observations during healing of a full-thickness human surgical wound by second intention. J Dermatol Surg Oncol. 1991 Dec;17(12):933-5. doi: 10.1111/j.1524-4725.1991.tb01692.x. PMID 1960262
- [Background] Zitelli JA. Wound healing by secondary intention. A cosmetic appraisal. J Am Acad Dermatol. 1983 Sep;9(3):407-15. doi: 10.1016/s0190-9622(83)70150-7. PMID 6630602
- [Background] Chern PL, Baum CL, Arpey CJ. Biologic dressings: current applications and limitations in dermatologic surgery. Dermatol Surg. 2009 Jun;35(6):891-906. doi: 10.1111/j.1524-4725.2009.01153.x. Epub 2009 Apr 6. PMID 19397669

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Started | 8 | 6
Completed | 7 | 4
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Includes all patients randomized to receive Porcine Xenograft or Second Intention healing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 75 [68.5 to 85.3] | 80 [70.3 to 82.3] | 78 [67.5 to 84.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Surgical Site [Count of Participants; unit: Participants]
  Shin | 4 | 0 | 4
  Calf | 0 | 2 | 2
  Ankle | 2 | 4 | 6
  Foot | 2 | 0 | 2
Initial post-op defect size, area (length x width) [Median (Inter-Quartile Range); unit: centimeters squared] | 5.7 [4.7 to 8.9] | 6.0 [3.2 to 10.7] | 5.7 [4.2 to 9.1]
Procedure type [Count of Participants; unit: Participants]
  Mohs | 8 | 5 | 13
  Excision | 0 | 1 | 1
Medication history: blood thinners [Count of Participants; unit: Participants] | 6 | 4 | 10
Medication history: immunosuppressants [Count of Participants; unit: Participants] | 0 | 1 | 1
Medication history: antibiotics [Count of Participants; unit: Participants] | 0 | 1 | 1
Medical history: Diabetes [Count of Participants; unit: Participants] | 4 | 1 | 5
Medical history: current tobacco use [Count of Participants; unit: Participants] | 0 | 0 | 0
Medical history: venous stasis [Count of Participants; unit: Participants] | 5 | 4 | 9
Medical history: Skin infection [Count of Participants; unit: Participants] | 0 | 1 | 1
Topical or systemic prophylaxis after surgery [Count of Participants; unit: Participants] | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS) Observer Scale Total Score
Description: The primary outcome will be the total score of the POSAS observer scale, assessed at the 3-month (+/- 1 month) follow-up visit by two blinded evaluators who will not be involved in the placement of the porcine xenograft. For each patient, scores from the two blinded investigators will be combined by calculating the mean. The POSAS (Patient and Observer Scar Assessment Scale) is a validated assessment tool used for the assessment of all types of scars by professionals and patients. The observer scale is comprised of 6 items (vascularity, pigmentation, thickness, relief, pliability, and surface area) scored on a scale from 1("like normal skin") to 10 ("worst scar imaginable"). The total score is calculated as the sum of the six items (range, 6-60).
Time Frame: Between 2.70 to 8.75 months
Population: The Modified Intention-to-Treat (mITT) Population consisted of all patients who received the study intervention and completed the 3-month office visit follow-up, during which the primary endpoint was evaluated.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 7 | 4
score on a scale | 17.0 [13.0 to 19.3] | 20.5 [20.0 to 20.6]
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney); An exact Wilcoxon two-sample test was performed owing to the small sample size and number of tied observations; Hodges-Lehmann median difference = -3.5, 95% CI 2-sided [-8.0 to -0.5] — Median difference is for Porcine Xenograft group minus No Porcine Xenograft group

2. Secondary Outcome: POSAS Patient Scale Total Score
Description: Study participants will complete the POSAS patient scale at the 3-month follow-up visit. The POSAS (Patient and Observer Scar Assessment Scale) patient scale consists of 6 items assessing patients' subjective opinion of scar quality in terms of pain, itching, color, pliability, thickness, and relief. Each item is scored from 1 (normal pigmentation, no itching, etc.) to 10 ("worst imaginable scar or sensation"). The total score of the POSAS patient scale is calculated as the sum of the six items (range, 6-60).
Time Frame: 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 7 | 4
score on a scale | 15.0 [13.0 to 17.5] | 18.0 [15.3 to 19.0]
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney); An exact Wilcoxon two-sample test was performed owing to the small sample size and number of tied observations; Hodges-Lehmann median difference = -2.5, 95% CI 2-sided [-9 to 12] — Median difference is for Porcine Xenograft minus No Porcine Xenograft

3. Secondary Outcome: Healing Time
Description: Healing time will be measured in weeks based on patient's responses to question 1 of the weekly follow-up questionnaire ("Is the wound completely healed (i.e., wound is completely closed with no open areas)?"). For example, a patient who first replies "Yes" to this question on the third weekly follow-up questionnaire will be assigned a healing time of 3 weeks. A more objective measure of healing time would not be feasible given our resources and patient schedule.
Time Frame: Up to 38 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 7 | 4
weeks | 14.0 [9.5 to 24.0] | 13.0 [9.25 to 20.25]
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney); An exact Wilcoxon two-sample test was performed owing to the small sample size and number of tied observations; Hodges-Lehmann median difference = 1.0, 95% CI 2-sided [-19.0 to 20.0] — Median difference is for Porcine Xenograft group minus No Porcine Xenograft group

4. Secondary Outcome: Ratio of Scar Size to Initial Defect Size
Description: The initial postoperative defect size will be measured by the investigator prior to intervention in terms of length and width using a sterile ruler. Initial defect area will be calculated as length times width. Scar size will be measured in terms of length and width at the 3-month follow-up visit, and scar area will be calculated as length times width. The outcome will be calculated by dividing the scar area by the initial defect area.
Time Frame: 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 7 | 4
ratio | 0.43 [0.31 to 0.54] | 0.35 [0.21 to 0.51]
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney); An exact Wilcoxon two-sample test was performed owing to the small sample size and number of tied observations; Hodges-Lehmann median difference = 0.01, 95% CI 2-sided [-0.26 to 0.33] — Median difference is for Porcine Xenograft vs. No Porcine Xenograft

5. Secondary Outcome: Pain Score at 1 Week Following Surgery
Description: Patients' pain scores will be measured based on their response to question 2 of the weekly follow-up questionnaire. Patients will be asked to rate their current pain level at the operative site on a scale from 1 (no pain) to 10 (worst imaginable pain).
Time Frame: 1 week
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 7 | 4
score on a scale | 1.0 [1.0 to 5.0] | 1.5 [1.0 to 3.3]
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney); An exact Wilcoxon two-sample test was performed owing to the small sample size and number of tied observations; Hodges-Lehmann median difference = 0, 95% CI 2-sided [-6 to 4] — Median difference is for Porcine Xenograft group minus No Porcine Xenograft group

6. Secondary Outcome: Number of Weeks With Pain Score Above 1
Description: as for outcome 5
Time Frame: 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 7 | 4
weeks | 2.0 [0.5 to 2.0] | 1.0 [0.75 to 1.25]
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); An exact Wilcoxon two-sample test was performed owing to the small sample size and number of tied observations; Hodges-Lehmann median difference = 0.5, 95% CI 2-sided [-1 to 2] — Median difference is for Porcine Xenograft group minus No Porcine Xenograft group

7. Secondary Outcome: Number of Participants With Infection
Description: Patient's charts will be reviewed at the completion of their 3-month office visit follow-up in order to analyze if they visited the dermatologist between the date of surgery and 3-month office visit and if infection was diagnosed.
Time Frame: 3 months
Population: The analysis population for this endpoint was the Safety Population, which consisted of all patients who receive the randomized study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 8 | 6
Participants | 2 | 2
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 1, Fisher Exact; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.03 to 13.3] — The "No Porcine Xenograft" group is the reference group

8. Secondary Outcome: Post-operative Bleeding Requiring Physician Intervention
Description: During each of the weekly follow-up questionnaires and during the 3-month follow-up visit, patients will be asked if they have experienced any post-operative bleeding that led to a visit to the physician (yes/no) and if there was any intervention performed by the physician to stop the bleeding (yes/no). The number and percentage of patients who experienced bleeding at any time during the 3-month follow-up period will be reported.
Time Frame: 3 months
Population: The analysis population for this outcome was the Safety Population, consisting of all patients who received the randomized study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 8 | 6
Participants | 0 | 1
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 0.43, Fisher Exact; Risk Difference (RD) = -0.167, 95% CI 2-sided [-0.564 to 0.185] — The risk difference is calculated as the outcome risk in the "Porcine Xenograft" group minus the outcome risk in the "No Porcine Xenograft" group. The confidence interval for the risk difference was calculated using the Newcombe hybrid score method

9. Secondary Outcome: Pain Score of 6 or Higher at One Week
Description: The proportion of patients with a pain score greater than or equal to 6 at the operative site will be assessed at one week following surgery. This will be based on the patient's response to the weekly follow-up questionnaire, with scores ranging from 1 (no pain) to 10 (worst imaginable pain).
Time Frame: 1 week
Population: The analysis population for this endpoint was all subjects in the Safety Population with a non-missing pain score at week 1. The safety Population consisted of all patients who received the randomized study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 8 | 5
Participants | 1 | 1
Statistical Analysis 1: Comparison: Porcine Xenograft Placement vs No Porcine Xenograft; Test type: Superiority; p = 1, Fisher Exact; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.006 to 55.9] — The "No Porcine Xenograft" group is the reference group

10. Post Hoc Outcome: Number of Patients Receiving Rescue Medication
Description: This outcome describes the number of patients in each treatment group receiving treatment with silver nitrate sticks as a "rescue medication" due to lack of complete wound healing at the 3-month (+- 1 month) visit following surgery.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
Number analyzed (Participants) | 7 | 4
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of the surgery until the patient's wound had completed healed as confirmed at a final follow-up visit. This timeframe ranged from approximately 3 months to 9 months.
Description: Adverse event data was collected during weekly phone interview with patients during the first 12 weeks of the study period. Adverse event data was also collected at the planned 3-month follow-up office visit and at subsequent office visits for patients who had not healed completely by 3 months.
Arm/Group | Porcine Xenograft Placement | No Porcine Xenograft
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 4/8 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Porcine Xenograft Placement (N=8) | No Porcine Xenograft (N=6)
Infection (Infections and infestations) | 2 (2) | 2 (2)
Post-operative Bleeding requiring intervention (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lymphedema drainage from wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-operative swelling, tenderness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stasis dermatitis flare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations include early termination due to discontinuation of the porcine xenograft product by the manufacturer, leading to small number of subjects analyzed. Primary outcome was assessed outside of the pre-planned follow-up window for several patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT03931746/Prot_SAP_000.pdf